CLINICAL TRIAL: NCT00334139
Title: A Prospective, Single-arm Multicenter Study to Evaluate Effect of Intravenous Zoledronic Acid on Bone Metabolism Given Over 4 Months in Patients With Prostate Cancer or Breast Cancer and Bone Metastasis
Brief Title: Effect of Zoledronic Acid on Bone Metabolism in Patients With Bone Metastasis and Prostate or Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EDE28
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Prostate Cancer; Breast Cancer; Bone Metastasis
Keywords: serum bone markers; bone metastasis; prostate cancer; breast cancer; quality of life; bisphosphonates
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- zoledronic acid (Experimental)
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — every 4 weeks for 4 months
  Other Names: ZOL446

SUMMARY:
Bisphosphonates have been used extensively in the treatment and the prevention of skeletal complications associated with bone metastases in patients with breast cancer and prostate cancer.

The purpose of this study is to assess the effect of zoledronic acid patients with prostate cancer or breast cancer and bone metastasis.

ELIGIBILITY:
Inclusion criteria:

* Prostate cancer with at least one cancer-related bone lesion with or without hormonal treatment.
* Breast cancer with at least one cancer-related bone lesion
* Negative pregnancy test at screening in case of child-bearing potential and Performance status ECOG 0-2
* Normal liver and kidney function
* Prior surgery, chemotherapy and radiotherapy is allowed. At least 4 weeks must have elapsed since the completion of surgery, chemotherapy and radiotherapy to breast or bone.

Exclusion criteria:

* Prior treatment with bisphosphonates within 6 months before study start, and during treatment with zoledronic acid. Known hypersensitivity to zoledronic acid or other bisphosphonates. Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L) or ≥12.0mg/dl (3.00 mmol/L)
* Current/active dental problems including
* infection of the teeth or jawbone
* dental or fixture trauma
* current or previous osteonecrosis of the jaw
* exposed bone in the mouth
* slow healing after dental procedures
* recent (within 6 weeks) or planned dental or jaw surgery (extraction, implants)
* Patients with clinically symptomatic brain metastases. Severe physical or psychological concomitant diseases expected to impair compliance with the provisions of the study protocol or impair the assessment of drug of patient safety
* Clinically significant ascites, NYHA III or IV, cardiac failure, clinically relevant pathologic findings in ECG
* History of diseases with influence on bone metabolism such as Paget´s disease and primary hyperparathyroidism and with need of treatment for osteoporosis (defined according to DVO, T-Score ≤2.5).
* Previous radiation therapy to bone (including therapeutic radioisotopes such as strontium 89) within 1 month

Additional protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Bone turnover assessed by bone turnover parameters | every 30 days

SECONDARY OUTCOMES:
Pain | every 30 days
Change in prostate specific antigen | every 30 days
Quality of Life | every 30 days
Correlation between pain and bone turnover | at end of study
Correlation between bone complications and bone turnover | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Ulm, Germany

REFERENCES:
- [Result] Thadepalli H, Gorbach SL, Broido PW, Norsen J, Nyhus L. Abdominal trauma, anaerobes, and antibiotics. Surg Gynecol Obstet. 1973 Aug;137(2):270-6. No abstract available. PMID 4723349